CLINICAL TRIAL: NCT03967717
Title: Correlation of Clinical and Laboratory Findings and Diuretic Efficacy in Patients With Edematous States in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Principal Investigator, University of Cologne
Other Study IDs: Protocol 1.0
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Edema
Keywords: Edema
MeSH Terms: conditions — Edema | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with edematous states: Patients with edematous states receive standard of care diuretic.
  Interventions: Other: Characterization of parameters of medical history, examination and diagnostics.

INTERVENTIONS:
Other: Characterization of parameters of medical history, examination and diagnostics. — Patients receive standard of care diuretics. The study only collects data to characterize parameters of medical history, examination and diagnostics.

SUMMARY:
The aim of the study is the characterization of parameters from medical history, physical examination and diagnostics, which correlate with and could be used to predict diuretic efficacy.

DETAILED DESCRIPTION:
This prospective observational study is conducted to identify and further isolate possible predictors for the efficacy of diuretics and to identify potential new predictors.

The study also observes if specific diuretic regimes (e.g. combination of loop diuretics and distal effective diuretics for sequential nephron blockade) have a greater diuretic effect. This is not yet proved.

The data of the study shall to help to determine criteria, allowing to choose an effective diuretic regime in different patient cohorts already at the beginning of therapy and to identify patients at high risk.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Edema (peripheral and/or pulmonal) of cardiac or renal genesis.

Exclusion Criteria:

* Persons who are in a dependency/employment relationship with the investigators.
* Accommodation in an institution by judicial or administrative order.
* Patients in need of ascites puncture and/or thoracentesis on admission day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of patients with edematous states of cardiac or renal genesis. Patients with liver cirrhosis and in need of ascites puncture and/or thoracentesis are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Multivariable regression analysis at 6±1 hours | 6±1 hours from timepoint of first diuretic administration in the emergency department
  Multivariable regression analysis at 6±1 hours from timepoint of first diuretic administration in the emergency department.
  Independent variables: diuretic dose, clinical characteristics, serum creatinine, serum urea, urine sodium, urine conductivity and others. The dependent variable will be urine volume 6±1h after diuretic therapy or the difference in weight before diuretic administration and 6±1 hours afterwards.
Multivariable regression analysis 24 hours time course | 24 hours time course from timepoint of first diuretic administration in the emergency departmentnistration
  Multivariable regression analysis over 24 hours time course from timepoint of first diuretic administration in the emergency department.
  Independent variables: diuretic dose, clinical characteristics, serum creatinine, serum urea, urine sodium, urine conductivity and others. The dependent variable will be urine volume at different timepoints (e.g. 6h, 18h, 24h) within a maximum of 24 hours after first diuretic administration

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided